CLINICAL TRIAL: NCT05474807
Title: Improving Employee Well-being Through an Internet-delivered Strengths Use Intervention: A Feasibility Study
Brief Title: Internet-delivered Strengths Use Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West University of Timisoara (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MEGSIS S3 Pilot
Record Dates: First submitted 2022-06-24; First posted 2022-07-26 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Burnout, Professional; Mental Health Wellness 1
Keywords: work engagement; burnout; employee wellbeing
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: One-armed study with baseline and post-intervention measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): The experimental arm will receive the online strengths use intervention program over a period of 6 weeks, through an LMS software solution.
  Interventions: Behavioral: Internet-delivered strengths use intervention

INTERVENTIONS:
Behavioral: Internet-delivered strengths use intervention — The online strengths use intervention program, will be based on Miglianico et al.'s (2020) general framework, following the theorized five stages: (1) preparation and commitment, (2) identification, (3) integration, (4) action, and (5) evaluation.
  As to increase participant engagement and motivation, gamification components will be embedded in several of these stages.
  The entire intervention will be delivered online via an LMS software solution.

SUMMARY:
The aim of the study will be to test the feasibility and acceptability of a novel online-delivered gamification-based intervention for the identification, development, and use of strengths in the organization. The program will be addressed to employees at the beginning of their careers and will have the aim of boosting their well-being and performance.

ELIGIBILITY:
Inclusion Criteria:

- participants should score 4.49 or lower (on a scale from 0 to 6) on work engagement;

Exclusion Criteria:

* workload which will impede following the intervention program (based on a filter Yes/No question);
* lack of internet access during the period of the implementation of the program (based on a filter Yes/No question).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Work engagement | Change from baseline to post-intervention (approximately 6 weeks).
  Work engagement will be measured with the Utrecht Work Engagement Scale (UWES-9). It has 9 items that form three dimensions, each with 3 items: vigor (e.g., "At my work, I feel bursting with energy"), dedication (e.g., "I am enthusiastic about my job"), and absorption (e.g., "I am immersed in my work"). This measure uses a 7-point agreement scale (0 = never, 6 = always).
Psychological capital (PsyCap) | Change from baseline to post-intervention (approximately 6 weeks).
  Psychological capital will be measured with the 12-item Psychological Capital Questionnaire. It has four subscales: hope ("At the moment, I feel quite fulfilled at work."), self-efficacy ("I feel confident presenting information to a group of colleagues."), resilience ("Usually, at work, I easily get over the stressful aspects."), and optimism ("I am optimistic about what will happen to me in the future regarding my job."). All 12-item are reported on a 6-point Likert scale (1 = strongly disagree, 6 = strongly agree).
Strengths use | Change from baseline to post-intervention (approximately 6 weeks).
  Strengths use will be measured with a set of six items, rated on a 0 (almost never) to 6 (almost always) Likert scale. A sample item is "I seek opportunities to do my work in a manner that best suits my strong points".

SECONDARY OUTCOMES:
Burnout | Change from baseline to post-intervention (approximately 6 weeks).
  Burnout will be assessed with the 12-item Burnout Assessment Tool (BAT). This questionnaire has four subscales: exhaustion (3 items; "At work, I feel mentally exhausted."), emotional impairment (3 items; "At work, I feel unable to control my emotions."), cognitive impairment (3 items; "At work, I have trouble staying focused.") and mental distance (3 items; "I struggle to find any enthusiasm for my work."). All items will be scored on a 5-point scale ranging from 1 (never) to 5 (always).
Job satisfaction | Change from baseline to post-intervention (approximately 6 weeks).
  Job satisfaction will be measured with the Michigan Organizational Assessment Questionnaire. The scale has three items with a response on a 7-point scale (1 = total disagreement, 7 = total agreement). A sample item reads: "In general, I like working here.".
Job performance | Change from baseline to post-intervention (approximately 6 weeks).
  Job performance will be assessed with a 7-item scale. Response options range on a Likert scale from 1 (strongly disagree) to 5 (strongly agree). A sample item is "I adequately complete my assigned duties.".
Positive affect | Change from baseline to post-intervention (approximately 6 weeks).
  Positive Affect (PA) will be measured with the 10 items of the Positive Affect Negative Affect Schedule (PANAS), representing different types of positive emotions (e.g., "excited", "inspired", and "enthusiastic"). Respondents will be asked to indicate to what extent they experienced these in the time frame of the intervention on a 5-point scale (1 = very slightly or not at all; 5 = very much).
Life satisfaction | Change from baseline to post-intervention (approximately 6 weeks).
  Life satisfaction will be measured with the five items of the Satisfaction with Life Scale. All answers are reported on a 7-point Likert scale (1 = totally disagree; 7 = totally agree); one item example being, "I am satisfied with my life".
Employability | Change from baseline to post-intervention (approximately 6 weeks).
  Employability will be measured with the four-item Perceived Employability Scale. Each item is rated on a 5-point liker scale (1 = totally disagree; 5 = totally agree). Higher scores represent higher levels of employability.

OTHER OUTCOMES:
Satisfaction with the intervention | At study completion (post-intervention), an average of 6 weeks.
  Satisfaction with the intervention will be measured using 22 items. We will use 6 items aiming at the program's content retrieved from a questionnaire used for measuring the alliance between trainers and trainees. The minimum score is 6 and the highest is 42. A higher score means a better outcome (increased satisfaction with the intervention). Also, we will use 16 items retrieved from a scale previously used for measuring the satisfaction with an online intervention. Nine of the items are measured on a Likert scale. The minimum score is 7 and the maximum is 42. A higher score means greater satisfaction. 7 items are open-ended questions.
System usability | At study completion (post-intervention), an average of 6 weeks.
  We will use a 10-item questionnaire designed to measure participants' satisfaction with the online platform used for the program delivery. The total score of the System Usability Scale ranges between 0 and 100. A higher score means a better outcome.
Treatment adherence | At study completion (post-intervention), an average of 6 weeks.
  The number of completed assignments; Quality of completed assignment (qualitative rating of the degree of completeness and depth of the answer for each assignment, conducted by two independent experts based on apriori established coding grids).

CONTACTS AND LOCATIONS:
Locations (1):
- West University of Timisoara, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bangor, A., Kortum, P. & Miller, J.A. (2009). Determining What Individual SUS Scores Mean: Adding an Adjective Rating Scale. Journal of Usability Studies, 4(3), 114-123.
- [Background] Camman, C., Fichman, M., Jenkins, D., & Klesh, J. (1979). The Michigan Organizational Assessment Questionnaire (University of Michigan, Ann Arbor, Michigan).
- [Background] Crawford JR, Henry JD. The positive and negative affect schedule (PANAS): construct validity, measurement properties and normative data in a large non-clinical sample. Br J Clin Psychol. 2004 Sep;43(Pt 3):245-65. doi: 10.1348/0144665031752934. PMID 15333231
- [Background] Luthans, F. L., Avolio, B. J., & Avey, J. A. (2007). Psychological Capital Questionnaire (PsyCap) [Database record]. APA PsycTests. https://doi.org/10.1037/t06483-000
- [Background] Schaufeli, W. B., Bakker, A. B., & Salanova, M. (2006). The measurement of work engagement with a short questionnaire: A cross-national study. Educational and psychological measurement, 66(4), 701-716. https://doi.org/10.1177/0013164405282471
- [Background] Schaufeli WB, Desart S, De Witte H. Burnout Assessment Tool (BAT)-Development, Validity, and Reliability. Int J Environ Res Public Health. 2020 Dec 18;17(24):9495. doi: 10.3390/ijerph17249495. PMID 33352940
- [Background] Tulbure BT, Rusu A, Sava FA, Salagean N, Farchione TJ. A Web-Based Transdiagnostic Intervention for Affective and Mood Disorders: Randomized Controlled Trial. JMIR Ment Health. 2018 May 24;5(2):e36. doi: 10.2196/mental.8901. PMID 29798831
- [Background] Van Woerkom, M., Mostert, K., Els, C., Bakker, A. B., De Beer, L., & Rothmann Jr, S. (2016). Strengths use and deficit correction in organizations: Development and validation of a questionnaire. European Journal of Work and Organizational Psychology, 25(6), 960-975. https://doi.org/10.1080/1359432X.2016.1193010
- [Background] Watson D, Clark LA. Negative affectivity: the disposition to experience aversive emotional states. Psychol Bull. 1984 Nov;96(3):465-90. No abstract available. PMID 6393179
- [Background] Williams, L. J., & Anderson, S. E. (1991). Job satisfaction and organizational commitment as predictors of organizational citizenship and in-role behaviors. Journal of management, 17(3), 601-617. https://doi.org/10.1177/014920639101700305
- [Background] Miglianico, M., Dubreuil, P., Miquelon, P., Bakker, A. B., & Martin-Krumm, C. (2020). Strength use in the workplace: a literature review. Journal of Happiness Studies, 21(2), 737-764. https://doi.org/10.1007/s10902-019-00095-w
- [Background] De Witte, H. (1992). Tussen optimisten en teruggetrokkenen. Een empirisch onderzoek naar het psychosociaal profiel van langdurig werklozen en deelnemers aan de Weer-Werkactie in Vlaanderen [Between optimists and withdrawns. An empirical investigation of the psychosocial profile of longterm unemployed and participants of the Back-to-Work Program in Flanders]. Leuven, Belgium: HIVA